CLINICAL TRIAL: NCT03387800
Title: A Randomized Controlled Trial Evaluating Efficacy of an Intervention Which Enhances Social Support and Positive Affect Through Online Social Networking in Smoking Cessations
Brief Title: RCT for Evaluation of Online Social Networking Intervention in Smoking Cessations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HMRF 1213049
Record Dates: First submitted 2017-12-18; First posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Self Efficacy; Health Behavior
Keywords: randomized controlled trial; smoking cessation; social support; positive effect; online social networking; theory-based
MeSH Terms: conditions — Health Behavior; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WeChat interactive peer support group (Experimental): Participants will be grouped together by the researcher to form closed online peer support groups (with group names they choose). Activities on the WeChat groups serve two functions: i) It enhances social support among peer members toward smoking cessation. ii) The online support group also enhances the participants' positive affect.
  Interventions: Behavioral: Basic health education messages; Behavioral: WeChat interactive peer support group
- Basic health education messages (Active Comparator): Members of the control group will receive health education messages that will also be sent to the intervention group through WeChat. The messages include topics on physical and psychological aspects of perceived severity of smoking and perceived benefits of smoking cessation, and tips/skills on resisting situational temptations that may lead to relapse.
  Interventions: Behavioral: Basic health education messages

INTERVENTIONS:
Behavioral: Basic health education messages — Messages containing basic health education materials, including perceived severity of smoking, perceived benefit of smoking cessation and tips on resisting situational temptations will be sent to the participants of both arms through WeChat after randomization takes place.
Behavioral: WeChat interactive peer support group — Participants will be grouped together by the researcher to form closed online peer support groups (with group names they choose). Activities on the WeChat groups serve two functions: i) It enhances social support among peer members toward smoking cessation. ii) The online support group also enhances the participants' positive affect.
  Arms: WeChat interactive peer support group

SUMMARY:
The proposed RCT evaluates the efficacy of the aforementioned novel 2-month online smoking cessation intervention in increasing 7-day point prevalence quit rate over a 6-month follow-up period among Chinese adult smokers in Hong Kong.

DETAILED DESCRIPTION:
Aims and hypothesis: The proposed RCT evaluates the efficacy of the aforementioned novel 2-month online smoking cessation intervention in increasing 7-day point prevalence quit rate over a 6-month follow-up period among Chinese adult smokers in Hong Kong. It is hypothesized that the quit rate of the intervention group would be higher than that of the control group at 6 month follow up (i.e. one-sided hypothesis).

Design and subjects: The RCT study will randomize participants into the intervention group or the control group. Prior to randomization, a baseline telephone survey will be conducted. Phone interviews will be conducted to evaluate the outcomes at Months 3 and 6 after completion of the intervention. Interviewers will be blinded from the randomization status. The inclusion criteria are: i) current smokers who have smoked at least one cigarette in the past seven days prior to the baseline survey, ii) age 18 years old or above, iii) able to communicate in Chinese (Cantonese), iv) having access to a smart phone or mobile electronic devices and social networking media (WeChat), v) willing to be followed up (Months 3 and 6), vi) should own a smart phone or a similar device.

Study instruments: Structured questionnaires.

Interventions: The 2-month intervention includes i) interactive online support groups and ii) immediate preventive 'SOS' cue to action messages to be sent to fellow support group members in need via WeChat. Besides, basic health education messages will be sent to both the intervention and the control groups.

Main outcome measures: self-reported 7-day point prevalence (pp) quit rate of smokers at 6 months post end-of-intervention.

Data analysis and expected results: Baseline characteristics between the two groups will be compared using t-test and chi-square test as appropriate. To evaluate efficacy in terms of the primary outcome, absolute risk reduction (ARR), relative risk reduction (RRR) and number needed to treat (NNT) at Months 3 and 6 and their 95% confidence intervals will be derived. Mixed effects models will be used to compare the differential changes on the outcome variables across the time points Months 0, 3 and 6 between the two study arms with adjustment for potential confounding variables. Significance differences in smoking cessation will be found among the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Current smokers who have smoked at least one cigarette in the past seven days prior to the baseline survey
* Age 18 years old or above
* Able to communicate in Chinese (Cantonese)
* Having access to a smart phone or mobile electronic devices and social networking media (WeChat), v) willing to be followed up (Months 3 and 6)
* Should own a smart phone or a similar device

Exclusion Criteria:

* Physically or mentally unfit
* Having participated in smoking cessation programs (last six months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-01-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported 7-day point prevalence (pp) quit rate | 6 months
  Self-reported 7-day point prevalence (pp) quit rate of smokers at 6 months post end-of-intervention

SECONDARY OUTCOMES:
Number of cigarettes consumed per day as compared to that of the baseline | 6 months
  Number of cigarettes consumed per day as compared to that of the baseline at 6 months post end-of-intervention
Positive and Negative Affect Scale score | 6 months
  Positive and Negative Affect Scale score as compared to that of the baseline at 6 months post end-of-intervention. Positive and Negative Affect Scale is consisted of two subscales, i.e. Positive Affect Scale (total score is ranged from 10 to 50, the higher value represents a better outcome) and Negative Affect Scale (total score is ranged from 10 to 50, the higher value represents a worse outcome). Two subscales will not be combined to compute a total score.
Smoking Self-Efficacy Questionnaire score | 6 months
  Smoking Self-Efficacy Questionnaire score as compared to that of the baseline at 6 months post end-of-intervention. The total score is ranged from 12 to 60. The higher values represents a better outcome.
Subjective Norms Scale score | 6 months
  Subjective Norms Scale score as compared to that of the baseline at 6 months post end-of-intervention. The total score is 6 to 30. The higher value represents a better outcome.
Attitude Towards Smoking Scale score | 6 months
  Attitude Towards Smoking Scale score as compared to that of the baseline at 6 months post end-of-intervention. The total score is ranged from 8 to 56. The higher values represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zixin Wang, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No